CLINICAL TRIAL: NCT02890199
Title: Effect of Local Anesthesia on Postoperative Pain Following Sacrospinous Ligament Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Collaborators: American Association of Gynecologic Laparoscopists (Other)
Responsible Party: Principal Investigator, Katie Propst, Fellow, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHC-2016-0169
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine group (Active Comparator): 0.5% lidocaine mixed with 1:200,000 epinephrine 70 milliliters (mL) will be used for local injection at the sacrospinous ligament and for anterior / posterior colporrhaphy
  Interventions: Drug: Lidocaine
- Bupivacaine liposomal group (Experimental): 1.3% bupivacaine liposomal (20 mL) injected at the sacrospinous ligament 0.5% lidocaine mixed with 1:200,000 epinephrine 50mL for the anterior / posterior colporrhaphy
  Interventions: Drug: Bupivacaine liposomal

INTERVENTIONS:
Drug: Bupivacaine liposomal
  Arms: Bupivacaine liposomal group
Drug: Lidocaine
  Arms: Lidocaine group

SUMMARY:
During surgery for pelvic organ prolapse, it is common for the surgeon to inject fluid into the vaginal tissues to help with tissue dissection. It is common that anesthetic medication is mixed into this fluid to help with pain control after surgery. Usually the pain medication injected is short-acting. In this study the investigators plan to compare the usual short-acting injected pain medication with a long-acting injected pain medication to evaluate whether this improves pain control after surgery.

One type surgical procedure for prolapse will be evaluated. The procedure is sacrospinous ligament fixation. This is suspension of the vagina to treat pelvic organ prolapse. Study participants will be randomized to one of two study groups:

1. Lidocaine group (short-acting medication).
2. Liposomal bupivacaine group (long-acting medication)

Information will be collected on study participants, including: demographics, procedure data, and post-operative information. The primary outcome of this study is determine if use of long-acting injected local anesthesia at the time of sacrospinous ligament fixation leads to less post-operative pain compared to short-acting local anesthesia.

Secondary outcomes include:

1. post-operative opioid medication use
2. return to baseline pain status
3. post-operative time to first bowel movement
4. post-operative antiemetic use (nausea medication)
5. results of voiding trial after surgery
6. patient satisfaction with pain control

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age ≥ 18 years, ≤95 years
3. Planned vaginal sacrospinous ligament fixation with anterior and/or posterior colporrhaphy (SSLF APC) to treat pelvic organ prolapse with or without retropubic mid urethral sling
4. Able to give informed consent to participate

Exclusion Criteria:

1. Male
2. Age <18 years, > 95 years
3. Unable or unwilling to give informed consent to participate
4. Pregnancy
5. History of chronic pelvic pain, narcotic abuse, or daily narcotic usage in the last six months
6. Known allergy / intolerance to either lidocaine, bupivacaine liposomal, ketorolac, motrin, or acetaminophen
7. Known renal or hepatic insufficiency
8. Planned hysterectomy at the time of prolapse repair
9. Planned transobturator mid urethral sling at the time of prolapse repair

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Visual analog pain scale | 1 to 120 hours post-operative
  post-operative pain

SECONDARY OUTCOMES:
Equivalents of morphine used for pain control post-operative while hospitalized | 1-2 days post-operative
  Post-operative opioid use, in hospital
Equivalents of morphine used from the time of hospital discharge to post-operative day 7 | 7 days post-operative
  Post-operative opioid use, after hospital discharge
Modified surgical pain scale | 3, 7, 14, 28 days post-operative
  Return to baseline pain status
Time to first bowel movement | 1-28 days post-operative
  Days to first postoperative bowel movement
Post-operative antiemetic use, in hospital | 1-2 days post-operative
Void trial | 1-2 days post-operative
  Results of in-hospital void trial
HCHAPS pain questionnaire | 48 hours post-operative
  Patient satisfaction with pain control

CONTACTS AND LOCATIONS:
Overall Officials: Katie Propst, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Urogynecology Division, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No